CLINICAL TRIAL: NCT01715584
Title: Is There an Adverse Drug Reaction Between Renin-Angiotensin System Blockade and Inhaled Anesthetics? - A Pilot Study. Optional Deoxyribo-Nucleic Acid Donation for the Study of Hypertension.
Brief Title: Is There an Adverse Drug Reaction Between Renin-Angiotensin System Blockade and Inhaled Anesthetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Craig Railton, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 5982
Record Dates: First submitted 2012-10-01; First posted 2012-10-29 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: Hypertension; Sevoflurane; Inhaled Anesthetic; Angiotensin Converting Enzyme Inhibitor; Angiotensin II Receptor Blocking Agent
MeSH Terms: conditions — Hypertension | interventions — Sevoflurane; Nitrous Oxide; Air; Nitrogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Angiotensin Converting Enzyme Exposed (Other): Sevoflurane/oxygen/air/nitrous oxide
  Hypertensive patients exposed to Angiotensin Converting Enzyme Inhibitors (ACE Inhibitors)will make up this arm.
  Preoperative Exposure to any of the following Angiotensin Converting Enzyme Inhibitors Enalapril (Vasotec/Renitec) Ramipril (Altace/Prilace/Ramace/Ramiwin/Triatec/Tritace) Quinapril (Accupril) Perindopril (Coversyl/Aceon) Lisinopril (Listril/Lopril/Novatec/Prinivil/Zestril) Benazepril (Lotensin) Imidapril (Tanatril) Zofenopril (Zofecard) Trandolapril (Mavik/Odrik/Gopten) Fosinopril (Fositen/Monopril)
  Interventions: Other: Sevoflurane/oxygen/air/nitrous oxide
- Angiotensin Receptor Blocker Exposed (Other): Sevoflurane/oxygen/air/nitrous oxide
  Hypertensive patients exposed to Angiotensin Receptor Blocking Agents (ARBs).
  Preoperative Exposure to any of the following Angiotensin II Receptor Blocking Agents Losartan(Cozaar) Candesartan (Atacand) Valsartan (Diovan) Irbesartan (Avapro) Telmisartan (Micardis) Eprosartan (Teveten) Olemisartan (Benicar) Azilsartan (Edarbi)
  Interventions: Other: Sevoflurane/oxygen/air/nitrous oxide
- Non ACE/ARB Exposed (Other): Sevoflurane/oxygen/air/nitrous oxide
  Hypertensive patients not exposed to angiotensin converting enzyme inhibitors or Angiotensin receptor blocking agents will be put into this arm.
  Interventions: Other: Sevoflurane/oxygen/air/nitrous oxide

INTERVENTIONS:
Other: Sevoflurane/oxygen/air/nitrous oxide — Patients in each arm will be randomized to receive either: 50 per cent oxygen, air, and sevoflurane or 50% nitrous oxide, oxygen and sevoflurane. They will then cross over to the other gas mixture. The depth of each the anesthetic will be varied from 0.8 MAC (minimum alveolar concentration) to 1.6 MAC in 0.2 MAC steps. Hemodyamic variables will be measured at each anesthetic concentration (average of five measurements). Time will be allowed for anesthetic agent equilibration. Paralysis and analgesia using rocuronium and fentanyl will be provided to ensure patients do not move at low (less than 1.0 MAC. It is estimated the time for the cross over experiment will be approximately six hours.
  Other Names: Sevoflurane (Sevorane, Ultane, Sojourn); 1,1,1,3,3,3-hexafluoro-2-(fluoromethoxy)propane; fluoromethyl hexafluoroisopropyl ether; Nitrous oxide; oxgyen; air; nitrogen

SUMMARY:
It is controversial whether or not patients whose Renin Angiotensin System is blocked for the treatment of hypertension suffer increased risk when undergoing surgery and anaesthesia.

The investigators wish to test the hypothesis: Blockade of the Renin Angiotensin System causes altered dose response under general anaesthesia in a dose dependant manner. The investigators wish to look for altered responses across the usual anaesthetic dosing range as measured by blood pressure and heart responses.

DETAILED DESCRIPTION:
There has been mixed results in retrospective studies examining the effects of renin angiotensin blockade for the treatment of cardiovascular disease and post operative outcomes. Studies done in high risk patients have shown increased risk of death if patients are exposed to angiotensin converting enzyme inhibitors and angiotensin blocking agents.

The hypothesis is that patients exposed to medications that block the renin angiotensin system have altered dose response (a type of adverse drug reaction) to inhaled anaesthetic agents in a dose dependant manner as measured by cardiovascular response, specifically systemic vascular resistance index.

This is a pilot study of hypertensive patients undergoing anaesthesia and composite head and neck surgery. The patients will be separated into three groups: Angiotensin converting enzyme inhibitor exposed, Angiotensin Receptor Blocking Agent exposed, and any other treated hypertension. Following separation into groups based upon preoperative medication exposures each group will be randomized to determine the order in which two types of inhaled anaesthetics are administered. Each subject will be randomized to receive either Sevoflurane/air/oxygen first or Sevoflurane/50 per cent nitrous oxide/oxygen second or vice versa. The dose of the anaesthetic will be adjusted across the dosing range from 0.8 MAC (minimum alveolar concentration) to 1.6 MAC in steps of 0.2 MAC.

Each subject will have hemodynamic parameters measured at each dose of anaesthetic at each MAC. Five measurements of hemodynamic parameters will be recorded to minimize the effects of surgery on each measurement. The hemodynamic variables will be measured using a Flotrak and Vigeleo monitor and the quantities to be measured are: heart rate, blood pressure, systemic vascular resistance, systemic vascular resistance index, cardiac output, cardiac index, central venous pressure, stroke volume variation.

The subjects are offered the opportunity to donate DNA for future study of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* age over 40
* composite head and neck tumor resection
* treated hypertension
* hypertension medications taken on morning of surgery (except diuretics)

Exclusion Criteria:

* patient refusal
* age less than 40 or over 80 years
* combined surgical procedures
* emergency surgery
* Left ventricular ejection fraction less than 50 per cent
* calculated creatinine clearance less than 60 mL per minute

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic Vascular Resistance Index (SVRI) | approximately every 5 minutes for 6 hours
  A calculated hemodyamic parameter that assesses the resistance the heart faces to the forward flow of blood. Corrected for body surface area. SVRI = (cardiac output/blood pressure)/body surface area.

SECONDARY OUTCOMES:
Heart Rate | approximately every 5 minutes for 6 hours
  number of heart beats per minute
Systolic Blood Pressure | approximately every 5 minutes for 6 hours
  force of blood flow (measured in mmHg)
Diastolic Blood Pressure | approximately every 5 minutes for 6 hours
  force of blood flow (measured in mmHg)
Central Venous Pressure | approximately every 5 minutes for 6 hours
  force of blood flow returning to the heart (measured in mmHg)
Cardiac Output (CO) | approximately every 5 minutes for 6 hours
  Calculated volume of blood flow in Litres per minute(measured in mmHg). Cardiac Output = mean arterial pressure/systemic vascular resistance.
Cardiac Index (CI) | approximately every 5 minutes for 6 hours
  Calculated volume of blood flow in Litres per minute(measured in mmHg/m2), corrected for body surface area. Cardiac Output = (mean arterial pressure/systemic vascular resistance)/body surface area.
Stroke Volume Varriation | approximately every 5 minutes for 6 hours
  Calculated variation in stroke volume between heart beats (blood pressure = stroke volume x rate x systemic vascular resisitance).measured in real time throughout experiment, and at each anesthetic concentration
Systemic Vascular Resistance | approximately every 5 minutes for 6 hours
  A calculated parameter reflecting the resistance the heart faces to the forward flow of blood. Not corrected for body surface area. SVR = cardiac ouptut / blood pressure. Measured at each concentraion of inhaled anesthetic

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Railton, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre - Victoria Campus, London, Ontario, Canada

REFERENCES:
- See also: Relevant Reference — http://www.ncbi.nlm.nih.gov/pubmed/20524103
- See also: Relevant Reference — http://www.ncbi.nlm.nih.gov/pubmed?term=J%20Am%20Coll%20Cardiol%202009%3B%2054%3A1778-84